CLINICAL TRIAL: NCT05784610
Title: Interest of the Automated Management of Deep Neuromuscular Blockade Monitoring : A Pilot Pre-post Quasi Experimental Study (CURATP)
Brief Title: Interest of the Automated Management of Deep Neuromuscular Blockade Monitoring (CURATP)
Acronym: CURATP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: CURATP; 2022-A01929-34 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2023-02-06; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Neuromuscular Blockade
Keywords: deep neuromuscular blockade; neuromuscular blockade monitoring; automated management; abdominal surgery; laparoscopy

STUDY DESIGN:
Intervention Model Description: Time 1: Non-automated neuromuscular blockade monitoring (TOF/PTC). As the NMB monitoring is depending on anesthesiologist usual practice and so only TOF measure is systematic, it is necessary to include a blind anesthesiologist measurement with the ATP mode in order to compare with data obtained during Time 2.
  Time 2: Automated neuromuscular blockade monitoring (ATP). TOF and PTC stimulations are regularly performed, and PTC is systematically performed if TOF = 0/4
Who Masked: Care Provider, Investigator
Masking Description: Masking only for the anesthesist in arms "Time 1"
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TOF/PTC (Active Comparator): Non-automated neuromuscular blockade monitoring (TOF/PTC). As the NMB monitoring is depending on anesthesiologist usual practice and so only TOF measure is systematic, it is necessary to include a blind anesthesiologist measurement with the ATP mode in order to compare with data obtained during Time 2.
  Interventions: Device: Monitorage by TOF/PTC; Device: Monitorage by ATP
- ATP (Experimental): Automated neuromuscular blockade monitoring (ATP). TOF and PTC stimulations are regularly performed, and PTC is systematically performed if TOF = 0/4. If PTC = 10/10, a TOF stimulation is automatically performed.
  Interventions: Device: Monitorage by ATP

INTERVENTIONS:
Device: Monitorage by TOF/PTC — Installation of TOFscan® and monitoring by MAR appreciation on one of the patient's wrists and installation of TOFscan® and monitoring by ATP mode (MAR blind) on the other wrist Installation of TOFscan® and monitoring by ATP mode
  Other Names: Installation of TOFscan®
  Arms: TOF/PTC
Device: Monitorage by ATP — Installation of TOFscan® and monitoring by ATP mode on one of the patient's wrists
  Other Names: Installation of TOFscan®

SUMMARY:
Neuromuscular blockade (NMB) recommendations updated in 2018 by the Société Française d'Anesthésie et Réanimation (SFAR) recommend the use of NMB agents to facilitate surgical procedure during abdominal surgery by laparotomy or laparoscopy.

This study aims to evaluate deep NMB monitoring with automated management of NMB depth measurement (ATP mode) versus non-automated monitoring (PTC/TOF), in order to improve the maintenance of deep NMB during abdominal surgery.

DETAILED DESCRIPTION:
The beneficial effects of deep NMB on the surgical conditions and thus the per and post operative surgical morbidity have been demonstrated in several studies, but the evidence are not yet consistent enough to make recommendations.

The monitoring of per operative NMB remains the rule, using the Train Of Four (TOF) at the ulnar nerve at the adductor of the thumb. However, when deep NMB for the most resistant muscles of the body is required (diaphragm and abdominal wall), the Post Tetanic Count (PTC) should be used.

In order to better adjust the NMB to the conditions of muscle relaxation required during surgery, an automatic mode called ATP for Automatic TOF/PTC has been developed (TofScan, Idmed, Marseille, France).

The investigators hypothesized that the use of the ATP would be able to better insure deep NMB, and to limit interventions on patients and/or on the NMB monitor during surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they meet all the following criteria :
* Age ≥ 18 years
* Scheduled Abdominal surgery by laparoscopy (digestive, urological and gynaecological) with a planned procedure duration of more than one hour, requiring deep NMB by rocuronium
* ASA I, II or III
* Free subject, without guardianship, curatorship or subordination
* Signed informed consent

Exclusion Criteria:

* Persons benefiting from enhanced protection, namely minors, persons deprived of their liberty by a judicial or administrative decision, adults under legal protection.
* Induction in rapid sequence,
* Use of an other NMB agent than rocuronium
* Predictable difficult intubation
* Persons participating in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Evaluate the monitoring of deep NMB by automated management of the measurement of depth NMB (ATP mode) compared to non-automated monitoring (PTC/TOF) in order to improve the maintenance of deep NMB during abdominal surgery | From intubation to surgical closure
  Percentage of time spent on deep NMB target during anesthesia, defined by PTC ≥ 1 and ≤ 5 responses

SECONDARY OUTCOMES:
Number of interventions by the anesthesia team to maintain deep curarization | From intubation to surgical closure
  Number of NMB agents reinjections and interventions on the NMB monitor by the anesthesia team, per hour, during the procedure
Amount of NMB agents administered | From intubation to surgical closure
  Total dose of NMB agents administered in mg/kg/h during the surgical procedure
Need to reverse NMB agents at the end of the procedure | From intubation to surgical closure
  Number of patients requiring NMB reversal with prostigmine or sugammadex
Effect of maintaining deep NMB at surgical level during the procedure | From intubation to surgical closure
  Maximum intra-abdominal pressure of insufflation in mmHg recorded during surgical procedure
Surgical conditions on the Leiden Surgical Rating Scale score | From intubation to surgical closure
  Surgical conditions will be measured using a translated French version of the Leiden Surgical Rating Scale ( L-SRS ), a likert scale from 1 "extremely poor conditions" to 5 "optimal conditions"

CONTACTS AND LOCATIONS:
Overall Officials: MATTHIEU M BOISSON, Professor, Principal Investigator — University Center Hospital of Poitiers
Locations (1):
- Centre Hospitalier de Poitiers, Poitiers, Vienne, France

REFERENCES:
- [Result] GRAY TC, HALTON J. Technique for the use of d-tubocurarine chloride with balanced anaesthesia. Br Med J. 1946 Aug 31;2:293-5. No abstract available. PMID 20996123
- [Result] Ali HH. A new device for monitoring force of thumb adduction. Br J Anaesth. 1970 Jan;42(1):83-5. doi: 10.1093/bja/42.1.83. No abstract available. PMID 4313564
- [Result] Dhonneur G, Kirov K, Motamed C, Amathieu R, Kamoun W, Slavov V, Ndoko SK. Post-tetanic count at adductor pollicis is a better indicator of early diaphragmatic recovery than train-of-four count at corrugator supercilii. Br J Anaesth. 2007 Sep;99(3):376-9. doi: 10.1093/bja/aem124. Epub 2007 Jun 7. PMID 17561516
- [Result] Kim HJ, Lee K, Park WK, Lee BR, Joo HM, Koh YW, Seo YW, Kim WS, Yoo YC. Deep neuromuscular block improves the surgical conditions for laryngeal microsurgery. Br J Anaesth. 2015 Dec;115(6):867-72. doi: 10.1093/bja/aev368. PMID 26582847
- [Result] Staehr-Rye AK, Rasmussen LS, Rosenberg J, Juul P, Lindekaer AL, Riber C, Gatke MR. Surgical space conditions during low-pressure laparoscopic cholecystectomy with deep versus moderate neuromuscular blockade: a randomized clinical study. Anesth Analg. 2014 Nov;119(5):1084-92. doi: 10.1213/ANE.0000000000000316. PMID 24977638
- [Result] Martini CH, Boon M, Bevers RF, Aarts LP, Dahan A. Evaluation of surgical conditions during laparoscopic surgery in patients with moderate vs deep neuromuscular block. Br J Anaesth. 2014 Mar;112(3):498-505. doi: 10.1093/bja/aet377. Epub 2013 Nov 15. PMID 24240315
- [Result] Madsen MV, Gatke MR, Springborg HH, Rosenberg J, Lund J, Istre O. Optimising abdominal space with deep neuromuscular blockade in gynaecologic laparoscopy--a randomised, blinded crossover study. Acta Anaesthesiol Scand. 2015 Apr;59(4):441-7. doi: 10.1111/aas.12493. Epub 2015 Mar 1. PMID 25789421
- [Result] Kim MH, Lee KY, Lee KY, Min BS, Yoo YC. Maintaining Optimal Surgical Conditions With Low Insufflation Pressures is Possible With Deep Neuromuscular Blockade During Laparoscopic Colorectal Surgery: A Prospective, Randomized, Double-Blind, Parallel-Group Clinical Trial. Medicine (Baltimore). 2016 Mar;95(9):e2920. doi: 10.1097/MD.0000000000002920. PMID 26945393
- [Result] Van Wijk RM, Watts RW, Ledowski T, Trochsler M, Moran JL, Arenas GW. Deep neuromuscular block reduces intra-abdominal pressure requirements during laparoscopic cholecystectomy: a prospective observational study. Acta Anaesthesiol Scand. 2015 Apr;59(4):434-40. doi: 10.1111/aas.12491. Epub 2015 Feb 13. PMID 25684372
- [Result] Koo BW, Oh AY, Seo KS, Han JW, Han HS, Yoon YS. Randomized Clinical Trial of Moderate Versus Deep Neuromuscular Block for Low-Pressure Pneumoperitoneum During Laparoscopic Cholecystectomy. World J Surg. 2016 Dec;40(12):2898-2903. doi: 10.1007/s00268-016-3633-8. PMID 27405749
- [Result] Yoo YC, Kim NY, Shin S, Choi YD, Hong JH, Kim CY, Park H, Bai SJ. The Intraocular Pressure under Deep versus Moderate Neuromuscular Blockade during Low-Pressure Robot Assisted Laparoscopic Radical Prostatectomy in a Randomized Trial. PLoS One. 2015 Aug 28;10(8):e0135412. doi: 10.1371/journal.pone.0135412. eCollection 2015. PMID 26317357
- [Result] Plaud B, Baillard C, Bourgain JL, Bouroche G, Desplanque L, Devys JM, Fletcher D, Fuchs-Buder T, Lebuffe G, Meistelman C, Motamed C, Raft J, Servin F, Sirieix D, Slim K, Velly L, Verdonk F, Debaene B. Guidelines on muscle relaxants and reversal in anaesthesia. Anaesth Crit Care Pain Med. 2020 Feb;39(1):125-142. doi: 10.1016/j.accpm.2020.01.005. Epub 2020 Jan 8. PMID 31926308
- [Result] Murphy GS, Szokol JW, Avram MJ, Greenberg SB, Shear TD, Deshur M, Benson J, Newmark RL, Maher CE. Comparison of the TOFscan and the TOF-Watch SX during Recovery of Neuromuscular Function. Anesthesiology. 2018 Nov;129(5):880-888. doi: 10.1097/ALN.0000000000002400. PMID 30130260
- [Result] Claudius C, Skovgaard LT, Viby-Mogensen J. Arm-to-arm variation when evaluating neuromuscular block: an analysis of the precision and the bias and agreement between arms when using mechanomyography or acceleromyography. Br J Anaesth. 2010 Sep;105(3):310-7. doi: 10.1093/bja/aeq162. Epub 2010 Jun 30. PMID 20595196